CLINICAL TRIAL: NCT03847363
Title: The Influence of Different Anesthesia and Postoperative Pain Management on Acute and Chronic Postsurgical Pain After Thoracic Surgery: a Prospective Study
Brief Title: The Influence of Different Anesthesia on Acute and Chronic Postsurgical Pain After Thoracic Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: cpsp-revisited
Record Dates: First submitted 2019-02-10; First posted 2019-02-20 (Actual); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Acute Pain; Chronic Postsurgical Pain
MeSH Terms: conditions — Acute Pain; Pain, Postoperative | interventions — Anesthesia, Epidural; Nerve Block

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- general anesthesia: patients underwent general anesthesia
- general and epidural anesthesia: patients underwent general and epidural anesthesia
  Interventions: Procedure: epidural anesthesia
- general anesthesia combined with nerve block: patients underwent general anesthesia combined with nerve block
  Interventions: Procedure: nerve block

INTERVENTIONS:
Procedure: epidural anesthesia — epidural anesthesia
  Groups: general and epidural anesthesia
Procedure: nerve block — paravertebral or serratus anterior plane block
  Groups: general anesthesia combined with nerve block

SUMMARY:
This study would compare acute and chronic postsurgical pain in patients underwent thoracic surgery with different anesthesia and analgesia methods, and explore the influencing factors.

DETAILED DESCRIPTION:
Chronic postsurgical pain (CPSP) was the pain caused by the operation that exceeded the healing time of normal tissue (usually 3 months), that was, a status that the damage caused by noxious stimulus had been healed, but the pain that cannot be explained by disease and inflammation were still existed. Due to the location of the incision and the necessity of indwelling the chest tube, the thoracic lung surgery was considered to be one of the most painful surgical operations. Studies have found that the incidences of CPSP in patients with thoracotomy were 57% (95% CI, 51-64%) and 47% (95% CI, 39-56%) at postoperative 3 and 6 months, respectively. With the development of minimally invasive techniques, thoracic surgery had gradually become less traumatic, and the number of surgical incisions was gradually developed into single port.Through ages, epidural analgesia with a combination of local anesthetics and opioids had long been considered the "gold standard" for postoperative analgesia in thoracic surgery. However, with the development of clinical anesthetics and the widespread use of nerve block techniques, it had been found that in open radical gastrectomy, there was no significant difference in the inhibition of intraoperative stress response between dexmedetomidine combined with general anesthesia and a combined general-epidural anesthesia. So, which anesthesia and analgesia method was "perfect" for a specific type of surgery procedure? This study would compare acute and chronic postsurgical pain in patients underwent different thoracic surgery procedure with different anesthesia and analgesia methods, and explore the influencing factors.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II
* underwent selective thoracic surgery

Exclusion Criteria:

* with severe cardiac, endocrine,immunologic or haematologic diseases
* medical history of chronic pain problems in chest area
* medical history of pain-relief or sedative medication
* not able to communicate with investigators

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: patients underwent selective thoracic surgery meeting inclusion and exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-07-30 (Estimated)

PRIMARY OUTCOMES:
numerical rating scale of acute postsurgical pain | at day1 post-operation
  numerical rating scale is a 11-point scale for patient self-reporting of pain, in which 0 stands for no pain and 10 stands for the most severe pain.
numerical rating scale of acute postsurgical pain | at day2 post-operation
  numerical rating scale is a 11-point scale for patient self-reporting of pain, in which 0 stands for no pain and 10 stands for the most severe pain.
numerical rating scale of chronic postsurgical pain | at 3rd month post-operation
  numerical rating scale is a 11-point scale for patient self-reporting of pain, in which 0 stands for no pain and 10 stands for the most severe pain.
numerical rating scale of chronic postsurgical pain | at 6th month post-operation
  numerical rating scale is a 11-point scale for patient self-reporting of pain, in which 0 stands for no pain and 10 stands for the most severe pain.

CONTACTS AND LOCATIONS:
Overall Officials: jing cang, Study Chair — Shanghai Zhongshan Hospital
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided